CLINICAL TRIAL: NCT04339010
Title: Effect of Hypopressive Gymnastics Associated or Not With Pelvic Floor Muscle Training in Women With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PT, Clinical Professor, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hypopressive gymnastics
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Urinary Incontinence; Quality of Life; Pelvic Floor Disorders
Keywords: Pelvic floor; Hypopressive exercise
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: This was a single-blind randomized controlled trial comparing the effect of AHT versus AHT associated with PFM contraction in incontinent women.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypopressive (Experimental): 1. st session: the meetings were provided by a physiotherapist, who also discussed the location and function of the pelvic organs, PFM, and the transversus abdominis (TrA) muscles. The participants learned how to activate TrA muscles. The training was performed during full expiration, the physiotherapist check and coordinate the group to maintain the Tra contraction. The women were also trained to inhale through the nose and exhale through the mouth maintaining an apical breathing pattern.
  2. nd session: The contractions were executed during six different positions the ones which they will keep following through the whole treatment.
  3. rd session: The patients were exposed to all the six positions (supplementary material) and their three variations (positions 1, 3, 5 and 6 ). Every meeting obeyed the same schedule through the five weeks of treatment and was accompanied by two physiotherapists.
  Interventions: Other: Hypopressive exercise
- Hypopressive + PFMC (Active Comparator): This group receives the same protocol than the Hypopressive group, but with a verbal command to realize the PFM contraction during the activation of the deep abdominal muscle.
  Interventions: Other: Hypopressive exercise; Other: Pelvic floor muscle contraction

INTERVENTIONS:
Other: Hypopressive exercise — The hypopressive exercise is performed mainly via transversus abdominis (Tra) activation. The exercise relaxes the diaphragm, decreases intra-abdominal pressure and may activate the abdominal and PFM simultaneously.
Other: Pelvic floor muscle contraction — Pelvic floor muscle contraction (PFMC) is performed through a sequence of contraction and relax the PFM. It will improve PFM strength and is effective for treating urinary incontinence.
  Arms: Hypopressive + PFMC

SUMMARY:
Aim: To verify the effects of the abdominal hypopressive technic (AHT) associate or not with pelvic floor muscle training (PFMT) in urinary incontinence (UI) symptoms and pelvic floor muscle strength. Methods: Randomized controlled trial. Thirteen incontinent women were randomly divided into an AHT group or AHT+PFMC group. Outcome assessment was carried out using digital palpation (modified Oxford grading scale), Peritron perineometer, and the International Consultation Incontinence Questionnaire-Short Form (ICIQ-SF) questionnaire. The treatment protocol consisted of five twice-weekly, 40-min one-on-one sessions. The participants were assessed only at baseline and after the intervention. Results: It is expected that the group who performed PFMC will improve the maximal voluntary contractions (MVC) and improve urinary incontinence symptoms, while the hypopressive exercise does not.

DETAILED DESCRIPTION:
This was a single-blind randomized controlled trial comparing the effect of AHT versus AHT associated with PFM contraction in incontinent women. The study was approved by the Research Ethics of Santa Catarina State University (number 3.712.850) and each participating provided the written informed consent signed. Women were randomly assigned to either an AHT group or the AHT associated with PFM contraction (AHT + PFMC) group. The first group underwent a hypopressive exercise program that does not stimulate the PFM contraction, while the other group receives the AHT associated with PFM contraction stimulated by the physiotherapist during the sessions. Following eligibility screening by the research, the women were allocated in an of the two groups. Group allocation results were concealed by opaque, sealed envelopes with serial numbers, and the participants were assigned at the second visit by opening envelops in a sequential manner, after their eligibility was assessed at the first visit. Study investigators were blinded to treatment allocation. Participants underwent a five weeks intervention after the first evaluation, and the final evaluation occurred one week later on a date according to the participant availability.

The first three sessions were designated to learn how to perform the exercises and your variations correctly were part of the five weeks intervention. The intervention was performed in a forty-minute training session in two-week meetings during five consecutive weeks. All women included in this trial, independently of the group, received standardized lifestyle advice including, when appropriate, instructions about weight loss, constipation, hydration and the avoidance of heavy lifting. It is very important to emphasize that the time dedicated to performing the daily exercises was similar. The therapist applying the protocol was appropriately trained especially for the trial and it was not the same professional who conducted the evaluations.

ELIGIBILITY:
Inclusion Criteria:18 years old and older, and having a complaint or diagnosis of urinary incontinence.

-

Exclusion Criteria: women will be excluded if they had diseases affecting the muscular and nerve tissues, chronic degenerative and/or cerebrovascular disease, or neurological conditions, or had previously undergone pelvic floor re-education programs. Besides that, only women with the ability to correctly contract their PFM proceeded to intervention.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence symptoms | Pre intervention and 1 week post intervention
  Will be assessed by evaluating the ICIQ-SF questionnaire that assesses the frequency, severity, and impact on the quality of life of urinary incontinence (UI). The three scored items of the ICIQ-UI SF are: [1] ''How often do you leak urine?'' (0 ''Never" 1 ''About once a week or less often,'' 2 ''Two or three times a week,'' 3 ''About once a day,'' 4 ''Several times a day,'' 5 ''All the time''), [2] ''How much urine do you usually leak?'' (0 ''None,'' 2 ''A small amount,'' 4 ''A moderate amount,'' and 6 ''A large amount''), and [3] ''Overall, how much does leaking urine interfere with your everyday life?'' (Visual analog scale ranging from 0 ''Not at all'' to 10 ''A great deal''). The answers result in a sum, with a minimum score of 0, and a maximum score of 21. Preliminary cut-off scores were set to 0 as ''continent status'' and 1 or more as ''incontinence status".

SECONDARY OUTCOMES:
Maximal voluntary contraction | Pre intervention and 1 week post intervention
  Peritron 9300® manometer will be used to assess the maximum voluntary contraction (MVC). An MVC of PFM will be asked to the participant and the peak value was recorded, this process was repeated 3 times. The mean value of these three pressure peaks corresponded to MVC of the PFM.
Vaginal resting pressure | Pre intervention and 1 week post intervention
  The Peritron manometer will be inserted into the vaginal canal and a rest period was given to control the influence of possible voluntary and involuntary contractions, in order to obtain the vaginal resting pressure measurement . The vaginal resting pressure value will be determined by the lowest pressure value during rest.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Health and Sport Sciences, Florianópolis, Santa Catarina, Brazil